CLINICAL TRIAL: NCT05909072
Title: The Boosting Effect of Hyaluronic Acid on Tranexamic Acid Microneedles in Melasma Patients: A Split- Face Study
Brief Title: Tranexamic Acid With Microneedling in Melasma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Norhan Anees, principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: melasma
Record Dates: First submitted 2023-02-17; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- right side of the face (Active Comparator): microneedling with tranexamic acid alone on the right side of the face
  Interventions: Drug: tranexamic acid microneedling
- Left side of the face (Active Comparator): microneedling with tranexamic acid combined with hyaluronic acid on the left side
  Interventions: Drug: Hyaluronic acid combined with tranexamic acid microneedling

INTERVENTIONS:
Drug: Hyaluronic acid combined with tranexamic acid microneedling — 1 ml of TXA, available as a 500 mg/5 ml ampoule, will be applied on the right side of the face after microneedeling and left to dry
  Arms: Left side of the face
Drug: tranexamic acid microneedling — On the left side of face, 0.5 ml of HA 3.5% will be used 1st followed by microneedling then 1 ml of TXA will be applied
  Arms: right side of the face

SUMMARY:
Topical tranexamic, a hydrophilic molecule, can't pass the lipid barriers of the stratum corneum and it's also not retained in adequate amount in the epidermis to enter the melanocytes, so there's a difficulty in the effective delivery of tranexamic acid into the melanocytes .

Hyaluronic acid was proved to improve the effective delivery of tranexamic acid through loosening corneocyte packing and helping TXA entering the melanocytes and minimizing its epidermal diffusion .

DETAILED DESCRIPTION:
Melasma is a common acquired pigmentary disorder characterized by irregular symmetric medium- to dark-brown macules and patches affecting the photoexposed areas of the face causing cosmetic disfigurement and low quality of life of the patient. Melsama affects mostly women of reproductive age with Fitzpatrick skin type IV-VI .

The exact pathogenesis of melasma isn't well-known, however the major etiological factors include genetic influences, chronic sun exposure, pregnancy, contraceptives, drugs and hormone therapy. Although the exact pathogenesis of melasma is not fully clarified, the pathophysiology of melasma is believed to involve excess production of melanin or an increase in the activity of melanocytes in the skin .

Melasma is often refractory to treatment with common relapses, so it needs a treatment modality that can be used for long time with minimal side effects. Topical depigmenting agents have good results but also may lead to many side effects.

Microneedling is a minimally invasive technique used for skin rejuvenation and treatment of many diseases, such as dyspigmentation. Gentle microneedling enhances upper dermal changes and increases the epidermal turnover that leads to decreasing melanin production and its deposition in melanocytes and also increasing the epidermal melanin cleareance which improve melasma.

Microneedling enhances transdermal drug delivery across the skin barrier through creating microchannels into the skin without causing actual epidermal damage. Microneedling with topical tranexamic acid (TXA) was proved to be safe, effective and comparatively painless without any detectable side effects.

Tranexamic acid, a hemostatic drug, is used to treat melasma by inhibiting the plasminogen activating system . The intracellular release of arachidonic acid, a precursor to prostaglandins E2, and the level of alpha-melanocyte-stimulating hormone increase as the result of plasmin activity. These two substances can activate melanogenesis. Therefore, the anti-plasmin activity of TA is thought as the main mechanism of hypopigmentory effect of this agent .

Tranexamic acid also inhibits angiogenesis of dermal blood vessels through suppression of vascular endothelial growth factor .

Topical tranexamic, a hydrophilic molecule, can't pass the lipid barriers of the stratum corneum and it's also not retained in adequate amount in the epidermis to enter the melanocytes, so there's a difficulty in the effective delivery of tranexamic acid into the melanocytes .

Hyaluronic acid (HA) was proved to improve the effective delivery of tranexamic acid through loosening corneocyte packing and helping TXA entering the melanocytes and minimizing its epidermal diffusion .

Hyaluronic acid also can actively adhere to melanocytes using cell suface HA receptors (such as cd44), so promotes the targeted delivery to melanocytes .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years.
* Both sexes.
* All types of melasma (epidermal, dermal and mixed).
* Nearly bilateral symmetrical melasma

Exclusion Criteria:

* Pregnancy and lactation
* Patients who are taking contraceptive pills at the time of the study or during the past 12 months.
* Patients with bleeding disorders with hypercoagulable state or the concomitant use of anticoagulants.
* Patient with history of thrombosis like DVT, coronary artery disease, stroke.
* Patient using any treatment for melasma during the past 1 month before the study.
* Active skin infection.
* Infection and immunosuppression
* Patient with keloidal tendency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Modified Melasma Area Severity Index (mMASI) score | through study completion, an average of 9 months
  Hemi-mMASI for each half of the face is calculated according to the following formula:
  Hemi-mMASI = 0.15 (A) (D) F + 0.3 (A) (D) M + 0.05 (A) (D) C
Physician global evaluation | through study completion, an average of 9 months
  The improvement of patients is evaluated regarding the improvement in mMASI ( ) and graded as follow:
  Poor (improvement < 25%) Fair (improvement 26%-50%) Good (improvement 51%-75%) Excellent (improvement >75%)
A five-point Likert scale for patient's satisfaction | through study completion, an average of 9 months
  Level of patient satisfaction is scored on five points:
  1. Not at all satisfied
  2. Not really satisfied
  3. Undecided
  4. Somewhat satisfied
  5. Very much satisfied
Pain assessment | through study completion, an average of 9 months
  Pain during the session will be assessed and graded as mild, moderate and severe
Dermoscopic evaluation | through study completion, an average of 9 months
  Dermoscopy will be performed for each patient at baseline, during and after each follow-up visit to evaluate the improvement of:
  * Color (light brown, brown, dark brown)
  * Pigmentation (pseudo network and arcuate lesions)
  * Vascularity (present or absent telangiectasia)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3800287/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4235096/
- See also: Related Info — https://bmcdermatol.biomedcentral.com/articles/10.1186/s12895-017-0066-5